CLINICAL TRIAL: NCT05824104
Title: Exploratory Study of Intermittent Hypoxia Treatment in Chronic Cerebral Hypoperfusion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, Principal Investigator, Capital Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IH-CCH
Record Dates: First submitted 2023-03-28; First posted 2023-04-21 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Chronic Cerebral Hypoperfusion

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients (Experimental): The intermittent hypoxia protocol refers to four cycles of 5 minutes hypoxia inhaling interval by 5 minutes normoxia, which is performed twice a day (at least 6 hours apart) in 7 days.
  Interventions: Other: Intermittent Hypoxia

INTERVENTIONS:
Other: Intermittent Hypoxia — The intermittent hypoxia protocol refers to four cycles of 5 minutes hypoxia inhaling interval by 5 minutes normoxia, which is performed twice a day (at least 6 hours apart) in 7 days.

SUMMARY:
This study aims to investigate the safety and efficacy of intermittent hypoxia treatment in patients with chronic cerebral hypoperfusion.

DETAILED DESCRIPTION:
Chronic cerebral hypoperfusion is a common and frequently occurring disease in middle-aged and senior people, and an important cause of multiple diseases such as acute ischemic stroke and vascular dementia. However, current treatments for chronic cerebral hypoperfusion are limited and nonspecific. Intermittent hypoxia refers to periodic intervention with alternating normoxia and hypoxia. Studies have shown that short-term (5-10min), low frequency (3-15 times), and mild to moderate hypoxia (9-16%) usually have protective effects and can improve cerebral blood perfusion. Therefore, this study is an exploratory study combining intermittent hypoxia treatment with chronic cerebral hypoperfusion, aiming to preliminarily explore the safety and potential effectiveness of intermittent hypoxia treatment in the using of chronic cerebral hypoperfusion.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 45-70 years, BMI 18.5-24kg/m2, both sexes.
* Subjects with risk factors of cerebrovascular disease, such as hypertension, diabetes, dyslipidemia, and so on, and the risk factors are well controlled.
* Cerebral/carotid ultrasound showed mild stenosis of unilateral internal carotid artery (ICA) or middle cerebral artery (MCA) (<50%) without stenosis of other major feeding arteries.
* Subjects with the manifestations of chronic cerebral hypoperfusion, such as dizziness, head pain, memory loss, slow reaction, inattention, emotional instability, decreased ability to work, sleep disorders and mood disorders, the course of more than 3 months.
* Subjects or their legally authorized representative can provide informed consent.

Exclusion Criteria:

* Stroke onset in the past 3 months, other severe neurological diseases, such as epilepsy, intracranial infectious diseases or demyelination.
* Uncontrolled hypertension (systolic blood pressure ≥200mmHg) with antihypertensive drugs before enrollment, other cardiovascular diseases.
* History of pulmonary, hepatic, dermatologic, or hematologic diseases.
* History of substance abuse.
* Pregnancy, hypertension, diabetes mellitus, obesity, sleep apnea and neurological disorders.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-05-10 (Estimated); Primary Completion 2023-09-10 (Estimated); Study Completion 2023-10-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse reactions | After the 7-day treatment.
  Adverse reactions included headache, vomiting, diarrhea, fatigue, dizziness (according to the Lake Louise scoring system), and insomnia.
Incidence of adverse reactions | Thirty days after the treatment.
  Adverse reactions included headache, vomiting, diarrhea, fatigue, dizziness (according to the Lake Louise scoring system), and insomnia.

SECONDARY OUTCOMES:
Tissue oxygen saturation | Baseline, after the 7-day treatment, 30 days after the treatment.
  Including peripheral oxygen saturation and brain tissue oxygen saturation (%).
Cerebral blood flow | Baseline, after the 7-day treatment.
  Cerebral blood flow will be detected by transcranial color-coded duplex sonography.
Neurobehavioral scale 1 | Baseline, after the 7-day treatment.
  It is evaluated by scales of Mini-mental State Examination (MMSE), which ranges from 0-30 points, and higher scores mean a worse outcome.
Blood pressure | Baseline, after the 7-day treatment, 30 days after the treatment.
  Including systolic blood pressure and diastolic blood pressure (mmHg).
Neurobehavioral scale 2 | Baseline, after the 7-day treatment.
  It is evaluated by scales of Montreal Cognitive Assessment (MoCA), which ranges from 0-30 points, and higher scores mean a worse outcome.

IPD SHARING:
Plan to Share IPD: No